CLINICAL TRIAL: NCT01038635
Title: Phase I/II Study of the Combination of 5-azacitidine With Lenalidomide in Patients With High Risk Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia (AML)
Brief Title: 5-Azacytidine With Lenalidomide in Patients With High Risk Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0467; NCI-2011-01941 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: 5-Azacytidine; 5-Aza; Lenalidomide; Revlimid; CC-5103; Myelodysplastic Syndrome; MDS; Acute Myelogenous Leukemia; AML
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Azacytidine + Lenalidomide (Experimental): 5-Azacytidine 75 mg/m^2 by vein daily x 5 days on days 1 to 5. Lenalidomide starting dose 10 mg orally daily x 5 days on days 6 to 10.
  Interventions: Drug: 5-Azacytidine; Drug: Lenalidomide

INTERVENTIONS:
Drug: 5-Azacytidine — 75 mg/m^2 IV daily x 5 days on days 1 to 5.
  Other Names: 5-AZA; Azacitidine; Vidaza; 5-AZC; AZA-CR; Ladakamycin
Drug: Lenalidomide — Starting dose 10 mg orally daily x 5 days on days 6 to 10.
  Other Names: CC-5013; Revlimid

SUMMARY:
The goal of Phase 1 of this clinical research study is to find the highest tolerable dose of lenalidomide that can be given in combination with azacitidine to patients with MDS or AML.

The goal of Phase 2 of this study is to learn if the combination dose of azacitidine and lenalidomide found in Phase 1 can help to control MDS and/or AML.

The safety of this drug combination will be studied in both Phases.

DETAILED DESCRIPTION:
The Study Drugs:

Azacitidine is designed to block certain proteins that stop the function of tumor-fighting genes. By blocking the "bad" proteins, the tumor-fighting genes may be able to work better.

Lenalidomide is designed to change the immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 6 groups of 3-6 participants will be enrolled in the Phase 1 portion of the study, and up to 40 participants will be enrolled in Phase 2.

If you are enrolled in the Phase 1 portion, the dose of lenalidomide you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of lenalidomide. Each new group will receive a higher dose of lenalidomide than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of lenalidomide is found.

If you are enrolled in the Phase 2 portion, you will receive lenalidomide at the highest dose that was tolerated in the Phase 1 portion.

All participants will receive the same dose level of azacitidine.

Study Drug Administration:

Each study "cycle" will be about 3-8 weeks, depending on how well you tolerate the drugs, any side effects that you may have, and how your blood count and bone marrow recovers.

On Days 1-5 of every cycle, you will receive azacitidine by vein over 15-30 minutes.

In order to participate in this study you must register into and follow the requirements of the Revlimid REMS™ program of Celgene Corporation. This program provides education and counseling on the risks of fetal exposure, blood clots and reduced blood counts. You will be required to receive counseling every 28 days during treatment with lenalidomide, follow the pregnancy testing and birth control requirements of the program that are appropriate for you and take telephone surveys regarding your compliance with the program.

If you are enrolled in Phase 2 of the study, on Days 6-15 of every cycle, you will take capsules of lenalidomide by mouth.

You should swallow lenalidomide capsules whole with a cup (about 8 ounces) of water at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose). If you take more than the prescribed dose of lenalidomide, you should seek emergency medical care if needed and contact study staff right away. Any unused lenalidomide should be returned as instructed through the RevAssist® program.

Any woman who can become pregnant should wear gloves if touching the lenalidomide capsules.

You have been informed of the risk of birth defects. If you are female, you agree not to become pregnant while taking lenalidomide. For this reason, lenalidomide is provided to patients under a special distribution program called Revlimid REMSTM.

Your dose of study drugs may be lowered if you experience side effects.

You may be given drugs to help prevent side effects, such as nausea, vomiting, and/or diarrhea. The doctor will tell you more about what drugs you may receive.

Study Visits:

At every study visit, you will be asked about any other drugs and/or treatments you may be receiving and about any side effects you may be having.

One (1) time during each week of Cycle 1:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.

On Days 21 and 28 of Cycle 1 (+/- 3 days), you will have a bone marrow aspiration performed to check the status of the disease. You will then have a bone marrow aspiration performed every 7-14 days for the rest of the study. If at any point the disease appears to go into remission, you will then have a bone marrow aspiration performed every 1-3 cycles.

Before Day 1 of Cycles 2 and beyond:

* Your medical history will be recorded.
* You will have a physical exam.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.

Pregnancy Testing:

If you are a woman who is able to become pregnant, you will have blood (about 1-2 tablespoons) or urine pregnancy tests 1 time a week for the first 4 weeks of the study, then every 4 weeks while on study, when you stop the study, and 4 weeks after you are off study.

If you are a woman who is able to become pregnant and your menstrual cycles are irregular, you will have blood (about 1-2 tablespoons) or urine pregnancy test 1 time a week for the first 4 weeks, then every 2 weeks while on study, when you stop the study, and 2 and 4 weeks after you are off study.

Length of Study:

You may continue to receive azacitidine as long as the doctor thinks it is in your best interest. You may receive lenalidomide as part of this study for as long as you are benefitting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

This is an investigational study. Both azacitidine and lenalidomide are FDA approved and commercially available for the treatment of MDS. Azacitidine is not FDA approved or commercially available for treatment of AML. The combination as used in this study is investigational.

Up to 88 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with higher risk MDS (bone marrow blasts >/= 10% to 30% inclusive) of any age who refuse or are not eligible for frontline chemotherapy.
2. No prior therapy for higher risk MDS as defined above.
3. Performance status of </= 2 by the Eastern Cooperative Oncology Group (ECOG) scale.
4. Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of University of Texas MD Anderson Cancer Center (UTMDACC).
5. Hydroxyurea for patients with rapidly proliferative disease can be used up to 24 hours prior to therapy but not concomitantly with 5-azacitidine or lenalidomide. Hydroxyurea can be used once the patient has completed the planned 5 azacitidine and lenalidomide treatment.
6. Adequate liver function: Total bilirubin of </= 1.5 x upper limit of normal (ULN), AST (SGOT) and ALT (SGPT) </= 3 x ULN
7. Renal function - assessed by calculated creatinine clearance as follows (see Appendix: Cockcroft-Gault estimation of CrCl): 1. Phase I subjects must have calculated creatinine clearance >/= 60ml/min by Cockcroft-Gault formula. 2. Phase II subjects must have calculated creatinine clearance >/= 30ml/min by Cockcroft-Gault formula.
8. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS®.
9. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
10. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
11. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
12. Continued from #9: Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

1. Nursing and pregnant females.
2. Known or suspected hypersensitivity to azacitidine or mannitol.
3. Patients with advanced malignant hepatic tumors.
4. Unwilling or unable to remain in compliance with the RevAssist® program
5. Known hypersensitivity to thalidomide or lenalidomide (if applicable).
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] DiNardo CD, Daver N, Jabbour E, Kadia T, Borthakur G, Konopleva M, Pemmaraju N, Yang H, Pierce S, Wierda W, Bueso-Ramos C, Patel KP, Cortes JE, Ravandi F, Kantarjian HM, Garcia-Manero G. Sequential azacitidine and lenalidomide in patients with high-risk myelodysplastic syndromes and acute myeloid leukaemia: a single-arm, phase 1/2 study. Lancet Haematol. 2015 Jan;2(1):e12-20. doi: 10.1016/S2352-3026(14)00026-X. Epub 2014 Dec 22. PMID 26687423
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 23, 2009 to June 21, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 94 participants registered, six were ineligible therefore not assigned to groups nor treated.
Groups:
- 5-AZA + LEN 10 mg: Phase I: 5-Azacytidine (5-AZA) + Lenalidomide (LEN): 5-Azacytidine 75 mg/m^2 by vein daily x 5 days on days 1 to 5 of each 28-day cycle. Lenalidomide starting dose 10 mg orally daily x 5 days on days 6 to 10.
- 5-AZA + LEN 15 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 15 mg orally for 5 days.
- 5-AZA + LEN 20 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 20 mg orally for 5 days.
- 5-AZA + LEN 25 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 25 mg orally for 5 days.
- 5-AZA + LEN 50 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 50 mg orally for 5 days.
- 5-AZA + LEN 75 mg for 5 Days: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 5 days.
- 5-AZA + LEN 75 mg for 10 Days: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 10 days.
- Phase II: AZA + LEN 50 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 50 mg orally for 10 days.
- Phase II: AZA+ LEN 25 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 25 mg daily for 5 days.
Period: Overall Study
Arm/Group | 5-AZA + LEN 10 mg | 5-AZA + LEN 15 mg | 5-AZA + LEN 20 mg | 5-AZA + LEN 25 mg | 5-AZA + LEN 50 mg | 5-AZA + LEN 75 mg for 5 Days | 5-AZA + LEN 75 mg for 10 Days | Phase II: AZA + LEN 50 mg | Phase II: AZA+ LEN 25 mg
Started | 5 | 3 | 3 | 3 | 4 | 3 | 7 | 20 | 40
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 15 | 38
Not Completed | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 2
Not completed — Disease Progression | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics represented in study phase, Phase I and Phase II separately.
Groups:
- 5-AZA + LEN 10 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 10 mg orally for 5 days
- 5-AZA + 50 LEN: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 50 mg orally for 5 days.
- 5-AZA + LEN 75 mg 5 Days: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 5 days.
- Phase II: 5-AZA + LEN 50 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 50 mg orally for 10 days.
- Total: Total of all reporting groups
Arm/Group | 5-AZA + LEN 10 mg | 5-AZA + LEN 15 mg | 5-AZA + LEN 20 mg | 5-AZA + LEN 25 mg | 5-AZA + 50 LEN | 5-AZA + LEN 75 mg 5 Days | 5-AZA + LEN 75 mg for 10 Days | Phase II: 5-AZA + LEN 50 mg | Phase II: AZA+ LEN 25 mg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 4 | 3 | 7 | 20 | 40 | 88
Age, Continuous [Median (Full Range); unit: years] | 65 [55 to 79] | 54 [54 to 66] | 66 [65 to 69] | 66 [54 to 71] | 71 [65 to 79] | 64 [63 to 77] | 63 [32 to 70] | 72 [36 to 88] | 66 [38 to 85] | 67 [32 to 88]
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 2 | 2 | 2 | 4 | 9 | 16 | 40
  Male | 4 | 2 | 0 | 1 | 2 | 1 | 3 | 11 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 4
  Not Hispanic or Latino | 4 | 3 | 3 | 2 | 4 | 3 | 6 | 18 | 37 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 6
  White | 5 | 2 | 3 | 3 | 4 | 2 | 5 | 18 | 36 | 78
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 3 | 3 | 4 | 3 | 7 | 20 | 40 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities for Determining Maximum Tolerated Dose (MTD) of Lenalidomide in Combination With 5-azacytidine (5-AZA)
Description: DLT determined only during first course of therapy, at least 28 days from treatment of last participant before a new dose level initiated. All severe (Grade 3-4) non-hematological toxicities that are drug related considered for DLT determination. If 1 participant develops grade III-IV non-hematological toxicity, 3 more will be accrued at that particular dose level. If 2 or more participants develop grade III-IV non-hematologic toxicity, the doses of the combination at which this occurs will be considered too toxic. A total of 10 patients will be treated at the maximally tolerated dose (MTD) of the combination (the dose level below that considered to be too toxic) to confirm its tolerability.
Time Frame: 3-8 week cycles, up to 24 weeks
Measure: Number; unit: participants
Groups:
- 5-AZA + 5 Days LEN 10 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 10 mg orally for 5 days.
- 5-AZA + 5 Days LEN 15 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 15 mg orally for 5 days.
- 5-AZA + 5 Days LEN 20 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 20 mg orally for 5 days.
- 5-AZA + 5 Days LEN 25 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 25 mg orally for 5 days.
- 5-AZA + 5 Days LEN 50 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 50 mg orally for 5 days.
- 5-AZA + 5 Days LEN 75 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 5 days.
- 5-AZA + 10 Days LEN 75 mg 75 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 10 days.
Arm/Group | 5-AZA + 5 Days LEN 10 mg | 5-AZA + 5 Days LEN 15 mg | 5-AZA + 5 Days LEN 20 mg | 5-AZA + 5 Days LEN 25 mg | 5-AZA + 5 Days LEN 50 mg | 5-AZA + 5 Days LEN 75 mg | 5-AZA + 10 Days LEN 75 mg 75 mg
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 4 | 3 | 7
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: 5-AZA + 5 Days LEN 10 mg vs 5-AZA + 5 Days LEN 15 mg vs 5-AZA + 5 Days LEN 20 mg vs 5-AZA + 5 Days LEN 25 mg vs 5-AZA + 5 Days LEN 50 mg vs 5-AZA + 5 Days LEN 75 mg vs 5-AZA + 10 Days LEN 75 mg 75 mg; Test type: Superiority or Other; Maximal tolerated dose = 75 — Maximal tolerated dose not reached as no dose limiting toxicity documented. MTD considered to be last dose level

2. Secondary Outcome: Overall Response Rate (ORR) of Lenalidomide in Combination With 5-azacytidine (5-AZA) in Participants With Leukemia
Description: Response defined as complete remission (CR) or complete remission with incomplete platelet recovery (CRi) for AML or any response for myelodysplastic syndrome (MDS) using international working group (IWG)-06 criteria. Complete response (CR) requires normalization of peripheral counts (absolute neutrophil count 10^9/L or more, platelet count 100 x 10^9/L or more), and a bone marrow with 5% or less marrow blasts. A hematologic improvement (HI) is defined as a CR with a platelet count above 30 x 10^9/L, without the need for transfusion of Platelets.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Phase I: 5-AZA + LEN MTD: 5-Azacytidine 75 mg/m^2 by vein daily x 5 days on days 1 to 5 of each 28-day cycle. Lenalidomide starting dose 10 mg orally daily x 5 days on days 6 to 10.
- Phase II: 5-AZA + LEN: All subjects received 75mg/m²/day AZA days 1-5 of each 28-day cycle. LEN 50 mg was administered orally for 10 days, with dose later amended to LEN 25 mg daily for 5 days.
Arm/Group | Phase I: 5-AZA + LEN MTD | Phase II: 5-AZA + LEN
Number analyzed (Participants) | 28 | 60
percentage of participants | 14 | 45

3. Secondary Outcome: Overall Response: Number of Participants With CR or CRi Response
Description: as for outcome 2
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Overall Study: 5-AZA + LEN MTD: Combined reporting for all phases, Phase I (5-Azacytidine 75 mg/m^2 by vein daily x 5 days on days 1 to 5 of each 28-day cycle. Lenalidomide starting dose 10 mg orally daily x 5 days on days 6 to 10) and Phase II All subjects received 75mg/m²/day AZA days 1-5 of each 28-day cycle. LEN 50 mg administered orally for 10 days, with dose later amended to LEN 25 mg daily for 5 days.
Arm/Group | Overall Study: 5-AZA + LEN MTD
Number analyzed (Participants) | 88
participants
  Complete Remission (CR) | 15
  Incomplete Count Recover (CRi) | 16

ADVERSE EVENTS:
Time Frame: Adverse events collected for 28 day cycle, up to 8 weeks following first course.
Groups:
- 5-AZA + LEN 10 mg: Phase I: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 10 mg orally for 5 days.
- 5-AZA + LEN 15 mg: Phase I: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 15 mg orally for 5 days.
- 5-AZA + 10 Days LEN 75 mg: 5-AZA 75 mg/m²/day Days 1-5 of each 28-day cycle + LEN 75 mg orally for 10 days.
Arm/Group | 5-AZA + LEN 10 mg | 5-AZA + LEN 15 mg | 5-AZA + LEN 20 mg | 5-AZA + LEN 25 mg | 5-AZA + LEN 50 mg | 5-AZA + 5 Days LEN 75 mg | 5-AZA + 10 Days LEN 75 mg | Phase II: AZA + LEN 50 mg | Phase II: AZA+ LEN 25 mg
Serious Adverse Events (participants affected / at risk) | 4/5 | 3/3 | 3/3 | 1/3 | 1/4 | 3/3 | 7/7 | 11/20 | 21/40
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 7/7 | 20/20 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-AZA + LEN 10 mg (N=5) | 5-AZA + LEN 15 mg (N=3) | 5-AZA + LEN 20 mg (N=3) | 5-AZA + LEN 25 mg (N=3) | 5-AZA + LEN 50 mg (N=4) | 5-AZA + 5 Days LEN 75 mg (N=3) | 5-AZA + 10 Days LEN 75 mg (N=7) | Phase II: AZA + LEN 50 mg (N=20) | Phase II: AZA+ LEN 25 mg (N=40)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Branchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-pulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyhydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage Central Nervous System (CNS) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infection other (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 4 (7) | 2 (2) | 3 (3)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 4 (6) | 6 (10)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Partial small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 3 (6)
Prolongation of hospitalization (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Right Femur Fracture (fall) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right Jaw Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombus (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5-AZA + LEN 10 mg (N=5) | 5-AZA + LEN 15 mg (N=3) | 5-AZA + LEN 20 mg (N=3) | 5-AZA + LEN 25 mg (N=3) | 5-AZA + LEN 50 mg (N=4) | 5-AZA + 5 Days LEN 75 mg (N=3) | 5-AZA + 10 Days LEN 75 mg (N=7) | Phase II: AZA + LEN 50 mg (N=20) | Phase II: AZA+ LEN 25 mg (N=40)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alteration in mental status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspergillus fungal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilateral parotitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
C. difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Change of smell (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain unclear etiology (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 16 (16)
Chronic obstructive pulmonary disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (caused chest pain) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatine Elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Infection, E-coli bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated bilirubin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcus bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 16 (16)
Fluid retention (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection/Skin nodules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Fungal pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 3 (3) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Gum Hemorrhage (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Gum infection (left jaw cellulitis and gingivitis) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0 (0)
influenzae, Haemophilus and stenotrophomonas (Infections and infestations) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0)
Hand tremors (Nervous system disorders) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Heart Palpitations (Cardiac disorders) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intracranial hemorrhage/bleed (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Jitteriness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Infection of intravenous line (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Macropapular rash on trunk (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7)
Night sweats (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-neutropenic fever (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
nonpruritic skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 10 (10)
possible chemotherapy-related cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 10 (10)
Renal failures (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0)
Scalp Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Severe muscle spasms of the lower back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendinitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subdural Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncopal Episode (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth Abcess/Infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Unsteady gait (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinarty Tract Infection (UTI) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vancomycin-resistant enterococci infection (VRE) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 8 (8) | 11 (11)
Pain, Right Flank (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes